CLINICAL TRIAL: NCT05052554
Title: Open-Label, Single-Dose, Exploratory Study With QR-504a to Evaluate Safety, Tolerability, and Corneal Endothelium Molecular Biomarker(s) in Subjects With Fuchs Endothelial Corneal Dystrophy With Trinucleotide Repeat Expansion in the TCF4 Gene (FECD3)
Brief Title: Study With QR-504a to Evaluate Safety, Tolerability & Corneal Endothelium Molecular Biomarker(s) in Subjects With FECD3
Acronym: Fuchs Focus
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No patients
Sponsor: ProQR Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PQ-504a-001
Record Dates: First submitted 2021-08-06; First posted 2021-09-22 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Fuchs Endothelial Corneal Dystrophy; FECD3; Corneal Diseases; LRS; Descemet's Membrane Disorder
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Corneal Diseases

STUDY DESIGN:
Intervention Model Description: QR-504a will be administered per intravitreal (IVT) injection, as a single dose. The starting dose is 30 µg. Guided by the dose (de-)escalation plan, doses in a range of below 30 µg and up to 60 µg may be evaluated following pre-specified criteria for opening additional dose cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30 µg cohort (Experimental): Open label single dose cohort: Dose level 1
  Interventions: Drug: QR-504a
- 60 µg cohort (Experimental): Open label single dose cohort: Dose level 2
  Interventions: Drug: QR-504a

INTERVENTIONS:
Drug: QR-504a — Intravitreal (IVT) injection

SUMMARY:
PQ-504a-001 (Fuchs Focus) is an open-label, single-dose, exploratory study to evaluate safety, tolerability, and corneal endothelium molecular biomarker(s) in subjects with Fuchs Endothelial Corneal Dystrophy with Trinucleotide Repeat Expansion in the TCF4 gene (FECD3).

DETAILED DESCRIPTION:
PQ-504a-001 (Fuchs Focus) is an open-label, intra-subject-controlled study in subjects with FECD3 scheduled for Descemet's Membrane Endothelial Keratoplasty (DMEK) in both eyes or with concurrent, preemptive lens replacement surgery (LRS/DMEK), if indicated as part of routine clinical practice. Each subject will go through the following two parts in this study:

• Part A without study drug administration: Part A of the study starts once LRS/DMEK of the first eye (hereafter called Eye 1) has been scheduled and subject eligibility has been confirmed. During the LRS/DMEK of Eye 1 corneal endothelium will be collected to assess the levels of selected molecular biomarkers. According to routine clinical practice, subjects will then be monitored for at least 4 weeks and up to approximately 6 months to evaluate recovery of Eye 1 prior to scheduling LRS/DMEK of the second eye (hereafter called Eye 2). The duration of the follow-up period also depends on the availability of cornea transplant material for Eye 2. Data generated during this part will serve as intra-subject control for data generated in Part B.

• Part B with study drug administration: Part B of the study starts once LRS/DMEK in Eye 2 can be scheduled and subject eligibility for Part B has been confirmed. At least 4 weeks prior to the scheduled LRS/DMEK in Eye 2, the subject will receive a single dose of QR-504a administered intravitreally in Eye 2. During the LRS/DMEK in Eye 2 corneal endothelium will be collected for molecular biomarker assessments and subjects will continue to be followed for safety and tolerability for at least 12 months post-surgery (ie, at least 13 months post dosing).

ELIGIBILITY:
Inclusion Criteria:

• Clinical diagnosis of FECD3 with:

* confirmed presence of trinucleotide repeat (TNR) expansion in the TCF4 gene (50 TNRs or more as determined by PCR),
* symmetrical disease progression in both eyes, in the opinion of the Investigator,
* a clinical indication for DMEK in both eyes ((phakic, aphakic, pseudophakic), or a clinical indication for concurrent, preemptive lens replacement surgery & DMEK in phakic eye.

Exclusion Criteria:

* Presence of any significant ocular or non-ocular disease/disorder which may either put the subject at risk because of participation in the study, may influence the results of the study, or the subject's ability to participate in the study.
* History of any form of keratoplasty in either eye.
* History or presence of ocular herpetic diseases (including herpes simplex virus, varicella zoster or cytomegalovirus) in either eye.
* Presence of any active ocular infection in either eye.
* Receipt within 3 months prior to Screening of in the opinion of the investigator any procedures or drugs that cause ocular disease or have ocular side effects that may confound assessment of safety, local tolerability or potential efficacy including.
* Systemic therapies known to influence the immune system (including but not limited to cytostatics, interferons, TNF-binding proteins, drugs acting on immunophilins, or antibodies with known impact on the immune system). Subjects that have been treated with systemic steroids within the past 12 months or that require intermittent use of topical steroids (eg, in pulmonological, dermatological or ophthalmological indications) may be considered for inclusion following approval by the Medical Monitor.
* Use of any investigational drug or device within 90 days or 5 half-lives of Day 1, whichever is longer, or plans to participate in another study of a drug or device during the study period.
* Any prior receipt of genetic or stem-cell therapy for ocular or non-ocular disease.
* Ongoing event of intraocular tumors.
* Pregnant or breastfeeding subjects. Female subjects of childbearing potential and male subjects must be sexually inactive by abstinence, which is consistent with the preferred and usual lifestyle of the subject, or agree to use highly effective methods of birth control, as defined in the study protocol. Women of non-childbearing potential may be included without the use of adequate birth control, provided the participant meets the criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of ocular and non-ocular adverse events (AEs) | 20 months
Change from baseline in the isoform levels of MBNL1 and MBNL2 in corneal endothelium | 20 months

CONTACTS AND LOCATIONS:
Overall Officials: ProQR Medical Monitor, Study Director — ProQR Therapeutics
Locations (1):
- Moorfields Eye Hospital, NIHR Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — http://www.proqr.com